CLINICAL TRIAL: NCT04358718
Title: Influence of Peri-operative Opioids on Circulating Tumor Cells in Patients Undergoing Robot-Assisted Laparoscopic Radical Cystectomy
Brief Title: Influence of Opioids on Circulating Tumor Cells in Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Principal Investigator, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CTC20200417
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer
Keywords: Circulating tumor cells; Opioid; Epidural anesthesia; Radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplastic Cells, Circulating | interventions — Anesthesia, General; Analgesia, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia (Active Comparator): Patients in this group will receive general anesthesia with intraoperative and postoperative intravenous opioid-based analgesia.
  Interventions: Procedure: general anesthesia
- general analgesia combined with epidural analgesia (Experimental): Patients in this group will receive combined epidural and general anesthesia with intraoperative and postoperative epidural ropivacaine-based analgesia.
  Interventions: Procedure: general anesthesia combined with epidural analgesia

INTERVENTIONS:
Procedure: general anesthesia — Patients will receive intraoperative and postoperative intravenous opioid-based analgesia for robot-assisted laparoscopic radical cystectomy.
  Arms: general anesthesia
Procedure: general anesthesia combined with epidural analgesia — Patients will receive epidural ropivacaine-based analgesia for robot-assisted laparoscopic radical cystectomy.
  Arms: general analgesia combined with epidural analgesia

SUMMARY:
Multiple lines of evidence have shown that perioperative opioids requirement was associated with poor outcomes in cancer patients, including increased cancer progression and metastases and reduced survival in patients with lung, breast, prostate, and bladder cancer. Circulating tumor cells (CTCs) have been validated as prognostic biomarkers of a number of cancers. The aim of this study is to investigate the effects of perioperative opioids on the number of CTCs in patients receiving robot-assisted laparoscopic radical cystectomy. The difference of the amounts of perioperative opioids is achieved by using general anesthesia combined with intravenous opioid-based analgesia intra- and post-operatively in one group and general analgesia combined with epidural ropivacaine-based analgesia in the other group.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* ASA I-II
* Patients with primary bladder cancer of Stage T2a or higher, who are scheduled for robot-assisted laparoscopic radical cystectomy
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Palliative surgery
* Contraindications for epidural anesthesia
* Metastatic bladder cancer
* Patients with a history of any other malignancy
* Chronic opioids medication
* severe systemic disease (heart, lung, kidney, or immune system)
* Known hypersensitivity or suspected allergy to intervention drugs
* Intellectual Disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
the number of circulating tumor cells | on the 3rd day after surgery
  The number of circulating tumor cells will be measured by collecting 5ml of venous blood sample.

SECONDARY OUTCOMES:
the number of circulating tumor cells | immediately after the surgery
  The number of circulating tumor cells will be measured by collecting 5ml of venous blood sample.
the number of circulating tumor cells | on the 30 day after surgery
  The number of circulating tumor cells will be measured by collecting 5ml of venous blood sample.
Visual Analogue Scale | at 24 hours after surgery
  Pain intensity will be assessed using the Visual Analogue Scale, which ranges from 0 to 10, with a higher score indicating greater pain intensity at 24 hours after surgery.
Visual Analogue Scale | at 48 hours after surgery
  Pain intensity will be assessed using the Visual Analogue Scale, which ranges from 0 to 10, with a higher score indicating greater pain intensity at 48 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Zhang S, Jin D, Luo J, Shi Y, Zhang Y, Wu L, Song Y, Su D, Pan Z, Chen H, Cao M, Yang C, Yu W, Tian J. mu-opioid receptor agonist facilitates circulating tumor cell formation in bladder cancer via the MOR/AKT/Slug pathway: a comprehensive study including randomized controlled trial. Cancer Commun (Lond). 2023 Mar;43(3):365-386. doi: 10.1002/cac2.12408. Epub 2023 Feb 5. PMID 36739595